CLINICAL TRIAL: NCT06990321
Title: A Single-center, Single-arm, Prospective Clinical Study of Intermediate-dose Cytarabine in Combination With Venetoclax for Consolidation Therapy of Middle- and High-risk Acute Myeloid Leukemia in The Elderly
Brief Title: Effectiveness of Medium-Dose Cytarabine Combined With Venetoclax for Consolidation Therapy in Elderly Patients With Intermediate to High-Risk Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yehui Tan (Other)
Responsible Party: Sponsor-Investigator, Yehui Tan, Professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-HS-084
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia (AML); Elderly
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Middle-and High-risk Acute Myeloid Leukemia in the Elderly (Experimental)
  Interventions: Drug: Intermediate-dose Cytarabine in Combination with Venetoclax

INTERVENTIONS:
Drug: Intermediate-dose Cytarabine in Combination with Venetoclax — Elderly patients with Middle- and High-risk Acute Myeloid Leukemia who received the Intermediate-dose Cytarabine in Combination with Venetoclax at the First Hospital of Jilin University from March 1, 2024 to December 31, 2026.

SUMMARY:
A Single-center, Single-arm, Prospective Clinical Study of Intermediate-dose Cytarabine in Combination with Venetoclax for Consolidation Therapy of Middle- and High-risk Acute Myeloid Leukemia in the Elderly

DETAILED DESCRIPTION:
This study is designed to be a prospective cohort study conducted at the First Hospital of Jilin University. The target populations of this study are patients with Middle- and High-risk Acute Myeloid Leukemia in the elderly who received intermediate-dose cytarabine in combination with venetoclax for consolidation therapy from June 1, 2025to December 31, 2026. It is expected to enroll 68 subjects in this study. The subjects' data such as demographics and other baseline characteristics, medications, prognosis, will be collected, and statistical analysis of data will be conducted to compare the effectiveness outcome measures

ELIGIBILITY:
Inclusion Criteria:

1.Age ≥ 60 years and ≤ 75 years, regardless of gender; 2.Diagnosed with AML (acute myeloid leukemia) according to WHO criteria (non-acute promyelocytic leukemia); 3.Risk stratification as intermediate or high risk based on the ELN (2022) guidelines; 4.Expected survival time ≥ 3 months; 5.Not suitable for allogeneic hematopoietic stem cell transplantation; 6.AML patients who achieve remission with morphologic assessment of bone marrow showing no leukemic involvement after induction therapy; 7.Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score of 0-2; 8.Meeting the following laboratory requirements (performed within 7 days prior to treatment):

1. Total bilirubin ≤ 1.5 times the upper limit of normal for the same age group;
2. AST and ALT ≤ 2.5 times the upper limit of normal for the same age group;
3. Serum creatinine < 2 times the upper limit of normal for the same age group;
4. Cardiac ejection fraction within normal limits as determined by echocardiogram. 9.Able to comply with the study visit schedule and understand and adhere to all trial protocol requirements; 10.Able to take oral medications.

Exclusion Criteria:

Subjects who meet any of the following criteria shall not be included in this study:

1. Allergic to any drugs included in the trial protocol or drugs with a chemical structure similar to the investigational drug.
2. Chemotherapy intolerance assessed by Ferrara 2013 criteria prior to enrollment.
3. Hematologic relapse (bone marrow blasts or immature cells exceed 5%).
4. Simultaneous diagnosis of other malignant tumors in organs (requiring treatment).
5. Known or suspected drug abuse or alcohol dependence.
6. Mental illness or any condition that prevents obtaining informed consent, or inability to comply with the study treatment and examination requirements.
7. Liver dysfunction (total bilirubin >1.5×ULN, ALT/AST >2.5×ULN, or liver-involved patients with ALT/AST >5×ULN), kidney dysfunction (serum creatinine >1.5×ULN).
8. Active heart disease, defined as one or more of the following:

1) History of uncontrolled or symptomatic angina. 2) Myocardial infarction within 6 months prior to enrollment. 3) History of arrhythmias requiring drug treatment or with severe clinical symptoms.

4) Uncontrolled or symptomatic congestive heart failure (>NYHA class 2). 5) Ejection fraction below the lower limit of normal. 9.Participation in another clinical trial within 30 days. 10.Active infection. 11.The investigator deems the subject unfit for participation in this trial.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival(RFS) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 36 months.
  Defined as the time from enrollment in this study to the occurrence of relapse. For patients without relapse, the time is calculated until death from any cause or the time of the last follow-up

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 36 months.
  Defined as the time from enrollment in this study to death from any cause. If the exact date of death is unknown, the time of death is defined as the last contact date. If the patient is still alive, the last observed time will be used, and the patient's OS will be considered for analysis.
Cumulative Relapse Rate (CIR) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 36 months.
  Defined as the proportion of patients who experience disease relapse from the time of enrollment in this study.
MRD Negative Conversion Rate | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 36 months.
  Defined as the proportion of patients who convert to MRD negative among all evaluable patients for efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China